CLINICAL TRIAL: NCT06649344
Title: A Phase III,Multicenter,Randomized,Open-label,Parallel-controlled Study Comparing the Efficacy and Safety of HRS9531 With Semaglutide in Subjects With Type 2 Diabetes Mellitus Not Adequately Controlled With Metformin Monotherapy or in Combination With SGLT2 Inhibitors
Brief Title: A Study of HRS9531 Versus Semaglutide Once Weekly as Add-on Therapy to Metformin Monotherapy or in Combination With SGLT2 Inhibitors in Participants With Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-303
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): HRS953-low dose
  Interventions: Drug: HRS9531 Injection
- Treatment group B (Experimental): HRS9531-high dose
  Interventions: Drug: HRS9531 Injection
- Treatment group C (Active Comparator): Semaglutide-1mg
  Interventions: Drug: Semaglutide Injection

INTERVENTIONS:
Drug: HRS9531 Injection — HRS9531 injected subcutaneously once weekly.
  Arms: Treatment group A; Treatment group B
Drug: Semaglutide Injection — Semaglutide injected subcutaneously once weekly.
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS9531 once weekly (QW) in subjects with type 2 diabetes mellitus not adequately controlled with metformin monotherapy or in combination with SGLT2 inhibitors compared to Semaglutide QW for 36 weeks and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes ≥ 90 days；
2. Stable daily dose(s) for ≥3months prior to screening of : 1) Any metformin formulations ≥1500 mg daily or maximum tolerated (≥1000mg daily). 2) Any metformin formulations ≥1500 mg daily or maximum tolerated (≥1000mg daily) with one type of SGLT-2 inhibitors;
3. Glycated hemoglobin was 7.5% ≤HbA1c ≤11.0%;
4. Female patients of childbearing potential and male patients must agree to use highly effective contraception during the trial and for at least 2 months after the last dose of the investigational medicinal drug. Female patients of childbearing potential must test negative for pregnancy at Visit 1 and not be breastfeeding.

Exclusion Criteria:

1. Known or suspected allergy or intolerance to the investigational medicinal products or related products；
2. Acute complications of diabetes occurred during the previous 6 months；
3. Serious chronic complications of diabetes in the past；
4. Use other antidiabetic drugs for ≥3months prior to screening ;
5. Before screening, have disease or treatment that may affect weight; or any previous condition that may affect gastric emptying； or gastrointestinal surgery;
6. Participation in any clinical trial of an approved or non-approved investigational product/treatment within the last 3 months or 5 half-lives, whichever is longer, prior to screening;
7. Any conditions that the Investigator judges might not be suitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 to Week 36
  Change from baseline in Glycosylated Haemoglobin after 36 weeks of treatment.

SECONDARY OUTCOMES:
Change in body weight | Week 0 to Week 36
  Change from baseline in body weight after 36 weeks of treatment.
Proportion of Subjects with HbA1c≤6.5% | Week 0 to Week 36
  Proportion of subjects with HbA1c≤6.5% after 36 weeks of treatment.
Proportion of Subjects with HbA1c<7% | Week 0 to Week 36
  Proportion of subjects with HbA1c<7% after 36 weeks of treatment.
Change in FPG (fasting plasma glucose) | Week 0 to Week 36
  Change from baseline in FPG after 36 weeks of treatment.
Change in FPG (fasting plasma glucose) | Week 0 to Week 52
  Change from baseline in FPG after 52 weeks of treatment.
7-points SMPG profiles | Week 0 to Week 36
  Fluctuation of 7-point SMPG. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner,120 minutes after start of dinner, before bedtime.
Incidence and severity of adverse events | Week 0 to Week 52+4 weeks follow-up
  Severity (mild, moderate and severe) is assessed by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhu Xianyi Memorial Hospital,Tianjin Medical University, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided